CLINICAL TRIAL: NCT03051061
Title: Effect of Antithrombotic Treatment in Patients With Both Coronary Heart Disease and Atrial Fibrillation:A Single-center,Retrospective,Observational Study
Brief Title: Effect of Antithrombotic Treatment in Patients With Both Coronary Heart Disease and Atrial Fibrillation
Acronym: ACHDAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Henan Institute of Cardiovascular Epidemiology (Other)
Responsible Party: Sponsor
Other Study IDs: HenanICE201604
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation; Coronary Heart Disease
Keywords: Atrial Fibrillation; Coronary Heart Disease; antithrombotic treatment; clinical prognosis
MeSH Terms: conditions — Atrial Fibrillation; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The optimal antithrombotic treatment for Coronary Heart disease (CHD) patients combined with Atrial Fibrillation (AF) is unresolved at present. Although the European and American guidelines have given a hand for us, there is absence of real-world data on the safety and efficacy of antithrombotic therapy in Asian populations. Only a few clinical trials are available to guide difficult decision on antithrombotic therapy in patients with combined AF and CHD，the investigators highlight the need for the rapid development of clinical trials to close the large gaps in evidence. This research aims to know the real-world use of antithrombotic treatment and clinical prognosis in Coronary Heart Disease patients complicated with Atrial Fibrillation.

DETAILED DESCRIPTION:
1. Our study is an observational, retrospective Study.
2. Key date elements and definition of each variable were in line with the American Heart Association(AHA)/European Society of Cardiology(ECS） recommendation on AF and CHD. To reflect the contemporary antithrombotic management of AF and CHD in the past five years, the following data were collected: basic socio-demographic information, symptoms and signs relating to AF, medical history, results of physical examination and laboratory test.
3. Follow-up time is at least 12 months. The patients will be asked about their medications and clinical outcomes by telephone interview or outpatient clinic. Then we will analyze the relative safety and efficacy of the various antithrombotic regimens.
4. Based on the largest prospective study by Denmark about this issue, we anticipate an 30% incidence of composite outcome in the triple therapy arm. To achieve a precision of 10% with an α=0.05 and the rate of defaulters is 10%. The final estimated sample size was 986.
5. Henan institute of cardiology epidemiology is responsible for design, date quality control and statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chest pain and a significant lesion >50% angiographically.
2. Patients with a documented AF as confirmed by 12 leads ECG or Holter ECG.

Exclusion Criteria:

1. Rheumatic valvular disease.
2. Contraindications to oral anticoagulation.
3. Combined with other serious diseases with a life expectancy < 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with coexisting coronary heart disease and atrial fibrillation
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2019-12-01 (Estimated)

PRIMARY OUTCOMES:
Thromboembolism | 1 year
  including ischemic stroke and systemic embolization

SECONDARY OUTCOMES:
Hemorrhage | 1 year
  according to GUSTO criteria
Major Adverse Cardiovascular Events(MACE) | 1 year
  death, congestive heart failure, myocardial infarction
A composite outcome | 1 year
  including thromboembolism,hemorrhage,all cause death,congestive heart failure, myocardial infarction

CONTACTS AND LOCATIONS:
Overall Officials: Changyu Gao, PhD, Principal Investigator — Henan Provincial People's Hospital; You Zhang, PhD, Principal Investigator — Henan Provincial People's Hospital; Lili Wei, MD, Principal Investigator — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No